CLINICAL TRIAL: NCT04130893
Title: Response of the Autonomic Nervous System to Auricular Stimulation of the Vagus Nerve (x)
Acronym: AURIX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator's decision
Sponsor: Hôpital Européen Marseille (Other)
Collaborators: Aix Marseille Université (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18-36
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2022-01

CONDITIONS: Vasoconstriction Disorder of Extremities
Keywords: ear acupuncture, auricular acupuncture

STUDY DESIGN:
Intervention Model Description: The study will consist of 3 sessions, It is a prospective crossover study. During the first session, the inclusion and non-inclusion criteria will be checked, then the cold water hand immersion test will be carried out to ensure the good tolerance of this test and then determine the basic values.
  During the second and third sessions, Two different auricular stimuli will be done to the ear during the hand immersion test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A stimulation of G13 then G15 (Experimental): The first session is similar between the two arms: Cold water hand immersion only At the Second session: Cold water hand immersion + G13 auricular stimulation At the Third session: Cold water hand immersion + G15 auricular stimulation
  Interventions: Behavioral: stimulation of G13 then G15
- B: stimulation of G15 then G13 (Experimental): The first session is similar between the two arms: Cold water hand immersion only At the Second session: Cold water hand immersion + G15 auricular stimulation At the Third session: Cold water hand immersion + G13 auricular stimulation
  Interventions: Behavioral: stimulation of G15 then G13

INTERVENTIONS:
Behavioral: stimulation of G13 then G15 — Study participant randomized into arm A will undergo a stimulation of point G13 at session N°2, then stimulation of point G15 at session N°3.
  Arms: A stimulation of G13 then G15
Behavioral: stimulation of G15 then G13 — Study participant randomized into arm B will undergo a stimulation of point G15 at session N°2, then stimulation of point G13 at session N°3.
  Arms: B: stimulation of G15 then G13

SUMMARY:
While invasive vagal stimulation has proven its therapeutic effectiveness over the past 20 years, particularly in the treatment of epilepsy or depression, its implementation is hampered by the high cost, high technicality and sometimes significant side effects. Non-invasive vagal stimulation, most often electric, is a less expensive therapeutic alternative and easier to implement, although the level of evidence is lower than that of invasive stimulation.

Some so-called traditional therapies, such as acupuncture, also stimulate certain parts of the ear by mechanical means, most often by puncturing the ear or the concha. In these traditional therapies, more than one hundred stimulation points have been described, each precisely positioned according to an empirical topography.

However, electrical non-invasive stimulation recognizes only three areas of interest on the ear, which are the areas of sensitive innervation, namely the afferences of the vagus nerve in the concha, which is the only one used in practice, the large occipital nerve on the lobe and part of the helix, and the auriculotemporal nerve on the rest of the auricular flag.

In this study, we would like to explore the justification for the topographic precision, adopted by traditional therapies, for non-invasive vagal stimulation on the concha.

DETAILED DESCRIPTION:
Main objective: to measure the physiological impact of two auricular stimuli on the same innervation territory but with opposite actions according to traditional therapies.

An identical physiological response on both stimulation points would be an argument against the topographical precision adopted by traditional therapies; conversely, a different physiological response would suggest the existence of a somatotopy nestled in the same innervation territory.

Secondary objectives:

* Determine, by sinus variability analysis, the intensity of the sympathetic and parasympathetic cardiac response of mechanical stimulation of the ear concha.
* Determine the existence of a blockage of the sympathetic reaction on cutaneous vasoconstriction after mechanical stimulation of the ear concha.
* Measure the relationship between sinus variability and paradoxical skin vasodilation after exposure to cold, as considered in the protocol.

To explore the justification for the topographical precision adopted by traditional therapies, we designed an experiment that consists of studying the autonomous, sympathetic and parasympathetic response to two stimuli performed over two different times.

The sympathetic stimulation will be done by immersing the right hand up to the wrist in a tub of cold water maintained at 5°C Mechanical parasympathetic stimulation will be performed on the ear in two different locations, by placing an adapted needle through an introducer to respect a standardized insertion depth.

The autonomous response will be measured by sinus variability, which responds to a double innervation, sympathetic and parasympathetic, and by the capillary skin response, which responds only to a sympathetic innervation.

The capillary skin response is measured by the amplitude and latency of the paradoxical vasodilation reflex following thermal stimulation, in this case the immersion of a limb's tip in cold water.

The study will consist of 3 sessions, as shown in the figure below. This is a prospective crossover study.

During the first session, the inclusion and non-inclusion criteria will be checked, then a water immersion test will be carried out to ensure the good tolerance of this test and then determine the basic values.

In the absence of acclimatization, the paradoxical vasodilation reflex is highly reproducible. During the second and third sessions, a mechanical stimulation will be done to the ear during the skin immersion test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, male and female, aged 18 to 60 years
* BMI (Body mass index) <=30
* Not participating in another clinical study with an investigational product

Exclusion Criteria:

* Drug treatment for cardiological, neurological or anticoagulant purposes
* History of diabetes, known neuropathy, high blood pressure, heart rhythm disorders, syncope or palpitation
* Known cryoglobulinemia
* Subject with Raynaud's syndrome
* Intra-auricular device of the piercing type,
* Psychoactive substance use, excessive alcohol consumption (>2 units per day chronically or >6 units per day recreationally) and tobacco (>5 cigarettes per day)
* Subject unable to read French
* Subject covered by Articles L1121-5 to 1121-8 of the Public Health Code, namely:
* Pregnant, postpartum and breastfeeding women
* Persons deprived of their liberty by a judicial or administrative decision
* Persons undergoing psychiatric care under Articles L3112-1 and L3113-1 who are not covered by the provisions of Article L1121-8
* Minors
* Persons of full age who are subject to a legal protection measure or who are unable to express their consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Skin temperature changes | 20 minutes
  measured by thermocouples placed on the following fingers: thumb, middle finger and ear of the right hand. The values and times of the minimum and maximum temperatures (latency and amplitude of (CIVD) Cold-Induced VasoDilatation waves) are measured

SECONDARY OUTCOMES:
Pain reported by the participant | 20 minutes
  Measured by visual analogue scale; this scale ranges from 0 to 10; 0 being no pain, 10 being excruciating pain.

OTHER OUTCOMES:
Sinus variability | 20 minutes
  measured by cardiofrequency meter(ACTIWAVE ®)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel SAGUI, MD, Principal Investigator — Hôpital Européen Marseille
Locations (1):
- Hôpital Européen Marseille, Marseille, PACA, France

REFERENCES:
- [Derived] Sagui E, Claverie D, Bidaut W, Grelot L. Heart rate variability and cold-induced vascular dilation after stimulation of two different areas of the ear: a prospective, single-blinded, randomized crossover study. BMC Complement Med Ther. 2024 Feb 13;24(1):83. doi: 10.1186/s12906-024-04392-7. PMID 38350937